CLINICAL TRIAL: NCT01102868
Title: An Randomized Controlled Trial of IMS-treatment Versus Scam for Canalis Carpi Syndrome
Brief Title: IMS-treatment and Canalis Carpi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMS1234
Record Dates: First submitted 2010-03-29; First posted 2010-04-13 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Needles

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Needle in acupuncture point Li11 (Sham Comparator): Acupuncture needle in the acupuncture point Li11
  Interventions: Device: Needle in acupuncture point Li11
- IMS of musculus pronator teres (Experimental): Acupuncture needle in musculus pronator teres
  Interventions: Device: IMS of the musculus pronator teres

INTERVENTIONS:
Device: Needle in acupuncture point Li11 — Acupuncture needle in acupuncture point Li11
  Other Names: Needles
  Arms: Needle in acupuncture point Li11
Device: IMS of the musculus pronator teres — Acupuncture needle in musculus pronator teres
  Other Names: Needles
  Arms: IMS of musculus pronator teres

SUMMARY:
Carpal tunnel syndrome is a condition in which the median nerve is compressed at the wrist, leading to paresthesias, numbness and muscle weakness in the hand. Treatment of the condition often involves surgery.

In this study we wish to se if there is an effect of using intramuscular stimulation (IMS) to release the tension of nervus medianus in the lower arm. The study will be performed by randomization to IMS of musculus pronator teres or a control ("Scam IMS treatment" to the acupuncture point Li11). The two insertion points are approximately 1cm apart in the lower arm.

DETAILED DESCRIPTION:
The most important outcome measure is ultra sound measured diameters for nervus medianus in the carpal tunnel

ELIGIBILITY:
Inclusion Criteria:

* Canalis Carpi Syndrome verified by ultrasound and clinically
* Both genders
* Age from 18 to 67

Exclusion Criteria:

* Negative neurophysiology result.
* Epilepsy,
* Heart disease,
* Rheumatism
* Unstable angina pectoris,
* Metal -allergy,
* Needle- phobia,
* Infection
* Hemophilia
* Cognitive problems

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Diameter of the Nervae medianus in the Carpal Tunnel | End 2011

SECONDARY OUTCOMES:
Health complaints | End 2011
Power of the hand grip | End 2011

CONTACTS AND LOCATIONS:
Overall Officials: Stein Atle Lie, Professor, Principal Investigator — Uni Health, University Research
Locations (1):
- Uni Health, Uni Research, Bergen, Norway

REFERENCES:
- [Derived] Kvist KB, Hilland R, Enehaug R, Schjelderup J, Lie SA, Halse AK. The treatment effect of intramuscular stimulation on carpal tunnel syndrome: A blinded randomized trial on 75 patients. J Bodyw Mov Ther. 2021 Jul;27:522-528. doi: 10.1016/j.jbmt.2021.03.020. Epub 2021 Apr 20. PMID 34391281